CLINICAL TRIAL: NCT02935439
Title: A Novel Fully Integrated Mobile Management Solution Using Cell Phone Technology for Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Principal Investigator, Stuti Dang MD, Clinical Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 20091057; 09KC-01 (Other Grant/Funding Number: James and Esther King Biomedical Research Program)
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Mobile Phone; Self-efficacy; Quality of Life; Knowledge; Feasibility
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell-Phone Intervention Arm (Active Comparator): A standard cell phone system sent web-browser messages daily to ask about their weight and symptoms of heart failure. Participants received up to 3 daily messages 15 minutes apart at a time of their choosing for 90 days. Participants were given a mobile phone for the 90 day period and a weight scale.
  Interventions: Other: Cell Phone
- Usual Care (No Intervention): Usual Care participants continued to receive care in the Heart Failure Clinic. All subjects were enrolled in the study for 90 days. Participants were given a weight scale.

INTERVENTIONS:
Other: Cell Phone — Participants responded to questions about their heart failure symptoms using a cell phone.
  Arms: Cell-Phone Intervention Arm

SUMMARY:
The purpose of this research study is to learn about the use of a cell phone for monitoring patients with heart failure. Participants will be asked questions about their heart failure daily and participants will need to answer them. The investigator will try to assess if the questions are easily understood by the participants. The investigator will also assess if the phone-based system for monitoring is easy to use by the participants. The investigator will also assess if the daily questions and interactions increase the self-efficacy, knowledge, and quality of life of participants related to their heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of heart failure
* Have an anticipated survival ≥ 6 months
* Receive care at the University of Miami or Jackson Healthcare system
* 18 years or older
* Able to communicate in English and/or Spanish
* Able to operate a cell phone, read, understand, and respond to the questions on the cell phone, and are able to use the weight scale.

Exclusion Criteria:

* Previous history of unstable coronary syndromes
* History of end-stage heart failure or heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease | 90 days
  This was used from the Chronic disease self-management program scales. (http://patienteducation.stanford.edu/research). Well-validated scale rating patient's confidence in managing chronic illness. It covers several areas of chronic diseases including symptom control, role functions, emotional functioning, and communicating with physicians. The English version has 6-items, while the Spanish version has 4-items.16 Using a Likert scale with item scores ranging from 1 to 10; scale score is the mean of the items.

SECONDARY OUTCOMES:
Health Distress Scale | 90 days
  This was used from the Chronic disease self-management program scales. (http://patienteducation.stanford.edu/research). Measures the distress associated with health problems over the last month. Using a Likert scale with item scores ranging from 0 to 5, scale score is the mean of the four items.
Communication with Physicians | 90 days
  This was used from the Chronic disease self-management program scales. (http://patienteducation.stanford.edu/research). Measures key behaviors to assess how well patients communicate with their healthcare providers. Using a Likert scale with item scores ranging from 0 to 5, scale score is the mean of the three items.
Fatigue Visual Numeric | 90 days
  This was used from the Chronic disease self-management program scales. (http://patienteducation.stanford.edu/research). Assesses self-reported fatigue in the past 2 weeks. This visual numeric scale is a modified version of the visual analog scale. It uses 10 bars of different heights and shading intensity.
Shortness of Breath Visual Numeric | 90 days
  This was used from the Chronic disease self-management program scales. (http://patienteducation.stanford.edu/research). Assesses self-reported shortness of breath in the past 2 weeks.
Heart Failure Self-Efficacy Scale-30 | 90 days
  30-item scale developed for self-efficacy with heart failure overall and with medications, diet, symptoms, activity, and heart failure readmission. Using a Likert scale with item scores ranging from 0 to 10, scale score is the mean of the items.
European Heart Failure Self-Care Behavior Scale | 90 days
  12-item questionnaire assesses self-care behavior of patients with heart failure. Using a Likert scale with item scores ranging from 1 to 5, scale score is the sum of responses.
Dutch Heart Failure Knowledge Scale | 90 days
  15-item questionnaire assesses heart failure knowledge in general, knowledge on heart failure treatment (including diet and fluid restriction) and heart failure symptoms and symptom recognition. Each correct answer gets one point and total score ranges from 0 to 15.
Minnesota Living with Heart Failure Questionnaire | 90 days
  21-item questionnaire assesses HF specific quality of life, using a 6-point Likert scale with item scores ranging from 0 to 5, scale score is the sum of responses.
The Medical Outcome Study 36-Item Short Form | 90 days
  36-item quality of life instrument used to evaluate perception of general health status, functional ability, and well-being.
Usability survey | 90 days
  31-item scale developed for this study to assess the participants' satisfaction with 7 aspects of the intervention using a 7-point Likert scale with item scores ranging from 1 to 7 (7 being best), and total score is the mean of responses. Patients were also asked open-ended questions in order to obtain an in-depth understanding of individual experiences, perceptions, concerns and feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Stuti Dang, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- Miami VA Healthcare System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No